CLINICAL TRIAL: NCT02309437
Title: Influences on the Nutrition Statuses and Clinical Outcomes of Early Use of Opioid to Control Local Mucosa Pain Induced by Irradiation in Nasopharyngeal Carcinoma Patients
Brief Title: Early Use of Opioid in Radiation Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PAIN-1
Record Dates: First submitted 2014-11-29; First posted 2014-12-05 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Nutrition Disorders; Quality of Life
Keywords: Nasopharyngeal carcinoma; Pain; Oxycodone; Opioids; Radiation mucositis
MeSH Terms: conditions — Nutrition Disorders; Nasopharyngeal Carcinoma; Pain | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild group (Experimental): Use oxycodone when pain is mild level. Start from 10 mg every 12 hours and titrate for appropriate dose.
  Interventions: Drug: Oxycodone
- Moderate group (Active Comparator): Use oxycodone when pain is moderate or severe level. Start from 10 mg every 12 hours and titrate for appropriate dose.
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Use oxycodone to treat patients with mild pain caused by radiation mucositis.
  Other Names: OxyContin
  Arms: Mild group
Drug: Oxycodone — Use oxycodone to treat patients with moderate/severe pain caused by radiation mucositis.
  Other Names: OxyContin
  Arms: Moderate group

SUMMARY:
This study is a superiority research to evaluate the safety and effectiveness of early use of oxycodone control release tablet for radiation mucositis in nasopharyngeal carcinoma patients.

DETAILED DESCRIPTION:
The present study is a prospective, randomizing, case-controlled, multi-center clinical trial. 174 firstly diagnosed nasopharyngeal carcinoma patients who need radical radiation therapy will be randomly divided into either early intervention or common intervention group. oxycodone control release tablets will be used to control the pain caused by radiation oral mucositis when the pain level is mild or moderate, respectively. The primary outcome measurement is nutrition status. Quality of life (QOL), the clinical outcomes, and the adverse effects are also to be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmed nasopharyngeal carcinoma;
2. Without historic chronic pain, no depend on analgesic drugs, no historic opioids intake;
3. Plan to receive radical radiation therapy, newly to radiation for head and neck;
4. Aged older or equal to 18 years old;
5. Could understand and cooperate to accomplish pain evaluation and observation scales;
6. Sufficient liver and kidney function: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) less than 2.5* upper limit of normal (ULN), serum creatinine less than 1.5*ULN;
7. Without other serious critical organ dysfunction, such as heart or lung dysfunction;
8. Performance status (PS) score less than 2;
9. Voluntary to participate and sign informed consent document;
10. Obey the rules of trail; could be followed-up on time.

Exclusion Criteria:

1. Excluded by inclusion criteria;
2. Known or suspected allergy to nonsteroidal anti-inflammatory drug (NSAID) or opioid medicine;
3. Unable to complete the follow-up;
4. Severe uncontrollable infections of medical disorders;
5. Major organ including heart, lung, kidney, or liver dysfunction;
6. With pathophysiological factors affecting drug absorption, distribution, metabolism or excretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Participants will be followed for the duration of radiotherapy, an expected average of 7 weeks.
  Body mass index (BMI, kg/m2) was defined as the body mass (kg) divided by the square of the body height (m).

SECONDARY OUTCOMES:
Numeric rating scale (NRS) | Participants will be followed for the duration of radiotherapy, an expected average of 7 weeks.
  NRS refers to the number 0-10 to indicate the degree of pain, 0 is painless and 10 is the most painful.
Hemoglobin | Participants will be followed for the duration of radiotherapy, an expected average of 7 weeks.
Albumin | Participants will be followed for the duration of radiotherapy, an expected average of 7 weeks.
Quality of life score | Participants will be followed for the duration of radiotherapy, an expected average of 7 weeks.
Dizziness | Participants will be followed for the duration of radiotherapy, an expected average of 7 weeks.
Nausea/vomiting | Participants will be followed for the duration of radiotherapy, an expected average of 7 weeks.
Somnolence | Participants will be followed for the duration of radiotherapy, an expected average of 7 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-ping Chen, M. D., Study Chair — Affiliated Cancer Hospital & Institute of Guangzhou Medical University; Bin Qi, M. D., Study Director — Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Locations (4):
- China (4):
  - Cancer Center Of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangzhou Panyu Center Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - People's Hospital of Boluo County, Huizhou, Guangdong

IPD SHARING:
Plan to Share IPD: No